CLINICAL TRIAL: NCT06697860
Title: Comparative Effect of Radial Shockwave Therapy and Graston Instrument Assisted Soft Tissue Mobilization on Plantar Fasciitis
Brief Title: Effect of Radial Shockwave Therapy and Graston Instrument Assisted Soft Tissue Mobilization on Plantar Fasciitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0112
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Plantar Fascia
Keywords: Radial Shockwave Therapy; Graston Instruments; Softtissue Mobilization; Plantar fascia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radial Shockwave Therapy (Experimental): Radial Shockwave therapy in Plantar Fasciitis.
  Interventions: Device: Radial Shockwave Therapy
- Graston instrument (Experimental): Graston Instrument assisted soft tissue mobilization on Plantar Fasciitis.
  Interventions: Device: Graston Instrument

INTERVENTIONS:
Device: Radial Shockwave Therapy — In Group A, Radial Shockwave Therapy (RST) was given to the plantar fascia for 5 minutes, with each session consisting of 5-10 shock wave pulses of varied intensity. Following that, stretching exercises for the plantar fascia and calf muscles were done for 30 minutes, with three sets of 30-second holds for each stretch. This therapy procedure was followed out in weekly sessions for 8 weeks, each lasting 40 minutes in total.
  Arms: Radial Shockwave Therapy
Device: Graston Instrument — Group B employed Graston Instrument-Assisted Soft Tissue Mobilization (IASTM) for 5-10 minutes to target and break down plantar fascia adhesions. The therapist used a specialized device to apply controlled, precise pressure to the fascia. Following that, stretching exercises for the plantar fascia and calf muscles were done for 30 minutes, with three sets of 30-second holds for each. The entire therapy procedure was carried out in weekly sessions for 8 weeks, each lasting 40 minutes in total..
  Arms: Graston instrument

SUMMARY:
Plantar fasciitis is a common musculoskeletal disorder characterized by inflammation of the plantar fascia, causing heel pain and discomfort. Various treatment modalities have been explored to alleviate symptoms, with Radial Shockwave Therapy (RST) and Graston Instrument-Assisted Soft Tissue Mobilization (IASTM) emerging as promising interventions.This study aims to compare the effectiveness of these two treatments in managing plantar fasciitis. RST offers a non-invasive alternative for individuals suffering from plantar fasciitis particularly crucial for patients who prefer conservative treatments or want to explore less invasive options before considering surgery also stimulate the body's natural healing processes by promoting blood flow and tissue regeneration.

DETAILED DESCRIPTION:
Study Design will be randomized clinical trial. Study setting will be Sehat medical complex Lahore. Study Duration will be 4 months after synopsis approval Sample size will be 40 calculated by Epitool ,intervention group will be Group A: Radial Shock Therapy(RST) , Group B: Graston Instrument Assisted Soft Tissue Mobilization (GIASTM). Purposive sampling technique will be implanted. Both genders (male/female).Age 20 to 45 years, Pre-diagnosed with chronic plantar fasciitis, Heel pain will be included. Patients with rheumatoid arthritis, osteoporosis and ankle and foot bursitis were excluded. VAS scale (visual analogue scale), Foot function index (FFI), 12-Item Short-Form Health Survey and goniometer will be data collection tools. SPSS version 25 will be used for statistical analysis. Shapiro-wilks test for normality will be used to assess the normality of the data after which it will be decided either parametric or non-parametric test will be used within and across the group.

ELIGIBILITY:
Inclusion Criteria:

* Both genders (male/female) Age 20 to 45 (25) unilateral chronic plantar fasciitis of more than 3 months Pre diagnosed with chronic plantar fasciitis soreness and local tenderness bottom of the heel. Searing or piercing type pain (26) Pain greater than four on the visual analogue scale (VAS) during the first steps in the morning(10) gradual development of pain with no trauma(27) pain generated by local pressure(26) Increase in pain in the morning upon taking a few steps or after prolonged non-weight bearing(28) symptoms decreasing with slight levels of activity, such as walking(11) No previous history of radial shockwave therapy or Graston technique for plantar fasciitis

Exclusion Criteria:

- Having lower limb pathology (24) Tarsal tunnel syndrome (TTS) Fat-pad syndrome(11) Have heel spurs(26) Bilateral PF Previous ankle or foot surgery History of topical corticosteroid injections to the ankle or foot Neuropathic or radicular pain in the lower limbs Participants with systemic diseases that cause foot discomfort, such as ankylosing spondylitis, osteoporosis psoriatic arthritis, rheumatoid arthritis, and gout, foot bursitis, as well as those with type I or type II diabetes and pregnancy, were also excluded from the study.(25)

Ages: 20 Weeks to 45 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-01-07 (Estimated); Study Completion 2025-01-07 (Estimated)

PRIMARY OUTCOMES:
Foot function Index | 8 weeks
  A Foot Function Index (FFI) was developed to measure the impact of foot pathology on function in terms of pain, disability and activity restriction. The FFI is a self-administered index consisting of 23 items divided into 3 sub-scales. Both total and sub-scale scores are produced. The FFI was examined for test-retest reliability, internal consistency, and construct and criterion validity. A total of 87 patients with rheumatoid arthritis were used in the study. Test-retest reliability of the FFI total and sub-scale scores ranged from 0.87 to 0.69. Internal consistency ranged from 0.96 to 0.73. With the exception of two items, factor analysis supported the construct validity of the total index and the sub-scales. Strong correlation between the FFI total and sub-scale scores and clinical measures of foot pathology supported the criterion validity of the index. The FFI should prove useful for both clinical and research purposes (29).
-Item Short-Form Health Survey | 8 weeks
  The 12-Item Short Form Health Survey (SF-12) was developed for the Medical Outcomes Study (MOS), a multi-year study of patients with chronic conditions. The resulting short-form survey instrument provides a solution to the problem faced by many investigators who must restrict survey length. The instrument was designed to reduce respondent burden while achieving minimum standards of precision for purposes of group comparisons involving multiple health dimensions. The instrument has been validated across a number of chronic diseases and conditions (22, 31-34) the test-retest reliability was found to be an ICC of 0.61 for PCS and 0.57 for MCS, adjusting for age, sex, race/ethnicity, and CRG.(31)
VAS (Visual analogue scale) | 8 weeks
  A Visual Analogue Scale (VAS) is one of the pain rating scale will be used for measuring the pain intensity with the categorization of none, mild, moderate and severe would suggest. It was to capture this idea of an underlying continuum that the VAS was devised (29) Reliability of VAS is high, ICC = 0.99 [95%CI 0.989 to 0.992] for 0 and 1 minute VAS scores. (30)
Goniometer | 8 weeks
  Goniometer: for measuring the ankle range of motion, goniometer will be used. Reliability of the goniometer was found for all measurements ranging from, Intra-class Correlation Coefficients for goniometry > 0.94. The concurrent validity of goniometer was good with ICC values of >0.85. The goniometer will be used to measure plantar flexion, dorsiflexion, inversion and eversion of the ankle joint.(35)

CONTACTS AND LOCATIONS:
Overall Officials: SABA RAFIQUE, MsPT(OMPT), Principal Investigator — Riphah International University
Locations (1):
- Sehat Medical Complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tu P. Heel Pain: Diagnosis and Management. Am Fam Physician. 2018 Jan 15;97(2):86-93. PMID 29365222
- [Background] Sichting F, Holowka NB, Ebrecht F, Lieberman DE. Evolutionary anatomy of the plantar aponeurosis in primates, including humans. J Anat. 2020 Jul;237(1):85-104. doi: 10.1111/joa.13173. Epub 2020 Feb 26. PMID 32103502
- [Background] Carek PJ, Edenfield KM, Michaudet C, Nicolette GW. Foot and Ankle Conditions: Plantar Fasciitis. FP Essent. 2018 Feb;465:11-17. PMID 29381040
- [Background] Yelverton C, Rama S, Zipfel B. Manual therapy interventions in the treatment of plantar fasciitis: A comparison of three approaches. Health SA. 2019 Sep 25;24:1244. doi: 10.4102/hsag.v24i0.1244. eCollection 2019. PMID 31934436